CLINICAL TRIAL: NCT00450099
Title: Determination of the Minimum Local Anesthetic Volume of 0.125% Bupivacaine in Labour Epidurals
Brief Title: Minimum Local Anesthetic Volume of Bupivacaine in Labour Epidurals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07-03; 05-0209-E
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Acute Pain
Keywords: Epidural; Labor Analgesia; Bupivacaine; Dose-response; Minimum effective volume
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Epidural, bupivacaine
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: bupivacaine — 0.125% bupivacaine in a volume determined according to the biased coin up-down sequential allocation model, starting at 8mL.

SUMMARY:
Different medications can be used as analgesics in labor epidurals. Bupivacaine is one of the most commonly used drugs for that purpose. The efficacy of a certain medication injected epidurally depends on the dose that is given. A certain dose can be administered in different concentrations, which will consequently mean different volumes. Our hypothesis is that for each concentration of a certain drug, there has to be a minimum effective volume that will be associated with the best possible performance of the drug. This study is being conducted to find the minimum volume of bupivacaine (a local anesthetic) that produces successful analgesia in 95% of patients in labor.

DETAILED DESCRIPTION:
Epidural administration of local anesthetics during labor produces analgesia, sympathetic block and motor block. The characteristics of the block depend on the volume and concentration of the local anesthetic that is used as well as the potential use of adjuncts. Although many researchers have investigated the efficacy of different drugs at different concentrations, the volumes used have been arbitrary. There is limited data regarding the minimum volume that is necessary for a successful anesthetic for a given concentration of bupivacaine.

This study is conducted as a prospective, randomized, up-down sequential allocation trial. The aim is to determine the minimum volume of 0.125% bupivacaine that will provide effective analgesia for 95% of parturients in the first stage of labor. The verbal numeric rating scale (VNRS) is used to rate the pain felt over the first 20 minutes, where 0 is no pain and 10 is the worst pain imaginable. After 20 minutes, if the VNRS was greater than 2, the volume of bupivacaine was considered inadequate and additional medication was given.

The volume of bupivacaine for the first patient was arbitrarily chosen as 8 ml, and the dose for each subsequent patient depends on the outcome of the previous injection. Doses will be increased or decreased in increments of 1 ml. If the previous response was ineffective, the next patient will receive 1 ml more than the last patient. If the response of the previous patient is effective, the Narayana rule, which is used to cluster doses around EV95, will be applied to determine if the dose remains the same or decreases.

50 patients will be included in the study. An estimate of EV95 will be calculated based on a logistic model with non-log-transformed doses, fit using Firth's penalized maximum likelihood approach for small sample bias correction. Confidence intervals will be calculated based on the profile likelihood approach.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Full term (more than 37 weeks gestation)
* Singleton pregnancy, vertex presentation
* Regular painful contractions occurring at least every 5 minutes
* Cervical dilatation < 5 cm

Exclusion Criteria:

* Any contraindication to epidural anesthesia
* Accidental dural puncture
* Allergy or hypersensitivity to bupivacaine
* Women who have received opioids or sedative medications within the last 4 hours

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Verbal Numeric Rating Scale (VNRS) less than or equal to 2 out of 10 during contraction | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada